CLINICAL TRIAL: NCT06712706
Title: Effect of Feeding Jejunostomy Placement on Sarcopenia in Patients with Advanced Stages of Esophageal Cancer in Curate Cancer Treatment
Brief Title: Effect of Feeding Jejunostomy on Sarcopenia in Patients with Esophageal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Stefan Gutknecht (Other)
Responsible Party: Sponsor-Investigator, Stefan Gutknecht, Principal Investigator, Stadtspital Zürich
Organization: Stadtspital Zürich (Other)
Other Study IDs: BASEC 2024-01793
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Esophageal Cancer; Esophageal Carcinoma; Sarcopenia; Feeding Tube
Keywords: feeding jejunostomy tube; enteral feeding route before or after neoadjuvant therapy; feeding jejunostomy tube at staging laparoscopy; feeding jejunostomy in esophagel cancer; sarcopenia in esophageal cancer; effect of enteral feeding on sarcopenia; sarcopenia in esophageal cancer patients
MeSH Terms: conditions — Esophageal Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with esophageal cancer receiving neoadjuvant therapy and an jejunal feeding tube: Included are:
  * Adult patients aged 18 years and above at the time of diagnosis.
  * Advanced-stage esophageal cancer or cancer of the esophageal junction and treated with curative intent, including neoadjuvant treatment.
  * Patients who received an FJT before neoadjuvant treatment or during definitive surgery.
  * Patients treated between 2017 and 2024 in the single institution of the City Hospital Zürich Triemli and completed 6 months of follow-up or died by 31.12.2024.
  Patients receiving the FJT at staging laparoscopy will be compared to patients receiving FJT at the time of esophagectomy.
  Interventions: Procedure: Feeding jejunostomy placement; Procedure: Feeding jejunostomy placement at esophagectomy

INTERVENTIONS:
Procedure: Feeding jejunostomy placement — Placement of feeding jejunostomy at staging laparoscopy
  Other Names: Early placement of FJT
Procedure: Feeding jejunostomy placement at esophagectomy — Placement of feeding jejunostomy at esophagectomy
  Other Names: Late placement of FJT

SUMMARY:
Participants were diagnosed with esophageal cancer needing chemo- or radiochemotherapy before the potentially curing surgery consisting of esophagectomy. At the time of diagnosis, in all participants, a laparoscopy to complete staging was performed. In some patients, a feeding jejunostomy tube (FJT) was placed at the time of staging laparoscopy; in others, the FJT was placed at the time of esophagectomy. A common risk factor for higher morbidity and mortality is sarcopenia, a condition associated with low skeletal muscle. This study aims to determine whether the timing of the FJT placement affects the progress of sarcopenia.

DETAILED DESCRIPTION:
At the City Hospital Zurich Triemli, an FJT tube is inserted in approximately two-thirds of patients before commencing neoadjuvant therapy. Another third receive an FJT at the time of esophagectomy to ensure postoperative enteral feeding. To this day, no prospective, randomized study exists as to whether placing an FJT at diagnosis or esophagectomy impacts sarcopenia. Retrospectively collected data is limited due to small sample sizes and observational character.

This is a retrospective, single-center cohort study using disease-related data already collected. The study design includes statistical balancing techniques to achieve comparability between the two groups and estimate an unbiased treatment effect of the timing of FJT placement.

All data is extracted from the clinical information systems and radiological systems and is credible, protected data. It is taken exclusively from the medical records; patients are not contacted for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years and above at the time of diagnosis.
* Advanced-stage esophageal cancer or cancer of the esophageal junction and treated with curative intent, including neoadjuvant treatment.
* Patients who received an FJT either before neoadjuvant treatment or during definitive surgery.

Exclusion Criteria:

* Insufficient data for analysis
* Written rejection of general consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated between 2017 and 2024 in the single institution of the City Hospital Zürich Triemli and completed a 6-month follow-up or died by 31.12.2024.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of the effect of timing of FJT placement on sarcopenia in patients with advanced stages of esophageal cancer in curative cancer treatment. | For each patient the investigated period is under one year. It starts with the time of diagnosis until approximately 6 months after esophagectomy.
  This will be measured by the skeletal muscle index (SMI) at three points: the first SMI is measured at the time of diagnosis, the second preoperatively at re-staging after completion of neoadjuvant therapy, and the third measurement is six months postoperatively.
  We expect that regular enteral feed through FJT during neoadjuvant therapy leads to higher SMI or less progress of sarcopenia compared to FJT placement at esophagectomy.

SECONDARY OUTCOMES:
Major complications | For each patient the investigated period is under one year. It starts with the time of diagnosis until approximately 6 months after esophagectomy.
  Classified according to Clavien-Dindo Classification and Comprehensive complication index, CCI.
Overall length of stay | For each patient the investigated period is under one year. It starts with the time of diagnosis until approximately 6 months after esophagectomy.
  The length of stay for esophagectomy and the overall length of hospital stay from diagnosis to six months postoperatively, excluding elective hospitalizations for radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Gutknecht, Dr. med., Principal Investigator — Stadtspital Zürich
Locations (1):
- Stadtspital Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No